CLINICAL TRIAL: NCT05025696
Title: Efficacy and Side Effects of Blacksoap® as Adjuvant Therapy of Scabies: a Single-blind Randomized Control Trial
Brief Title: Efficacy and Side Effects of Blacksoap® as Adjuvant Therapy of Scabies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Sandra Widaty, SpKK (K), Senior Lecturer, Department of Dermatology Venereology, Faculty of Medicine Universitas Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-08-0966
Record Dates: First submitted 2021-08-13; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies

STUDY DESIGN:
Intervention Model Description: A random cluster sampling was done on the population member diagnosed with scabies based on the boarding school building location into the intervention group and control group. The intervention group was receiving permethrin 5% cream and Blacksoap®, while the control group was receiving permethrin 5% cream and baby soap.
Who Masked: Investigator
Masking Description: The investigators who scraped the skin and did the transepidermal water loss examination were blinded on which arm the subjects were allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Blacksoap(R) applied whole body twice daily
  Interventions: Other: Blacksoap(R)
- Control (Placebo Comparator): Johnson and Johnsons Baby Soap applied whole body twice daily
  Interventions: Other: Blacksoap(R)

INTERVENTIONS:
Other: Blacksoap(R) — Blacksoap(R)

SUMMARY:
Background: Scabies is a skin disease due to Sarcoptes scabiei. The transmission risk is high among communities living together, such as dormitories, boarding schools, nursing homes, and so on. Blacksoap® is a soap product that is recognized as adjuvant therapy. Until now, there has been no research on the effectiveness and side effects of using Blacksoap®. Purpose: This research aimed to assess the cure rate of standard scabies treatment, with and without Blacksoap®, to determine pruritus visual analog scale (VAS) score, transepidermal water loss (TEWL) score before and after receiving therapy, and to evaluate the side effects of the treatment. Methods: The intervention group obtained standard therapy and Blacksoap®; meanwhile, the control group received standard therapy and baby soap.

DETAILED DESCRIPTION:
This study is a single-blind randomized clinical trial on scabies patient population at Pondok Pesantren Al Islami, Cibinong, Bogor. It is part of a research and social service by the Dermatology and Venereology Department of Faculty of Medicine Universitas Indonesia / dr. Cipto Mangunkusumo National Central General Hospital entitled "Early Detection of Scabies and Other Dermatoses and Evaluation of Scabies Treatment in Al-Hidayah and Al Islami Islamic Boarding School" Research subjects who are participating are those diagnosed with scabies (fulfilling 2 out of 4 cardinal signs of scabies).

The research was conducted from September to October 2018 with the entire scabies patient in Indonesia as the target population, and all students at Al Islami Boarding School who at the time had scabies as the accessible population. A random cluster sampling was done on the population member diagnosed with scabies based on the boarding school building location into the intervention group and control group. The intervention group was receiving permethrin 5% cream and Blacksoap®, while the control group was receiving permethrin 5% cream and baby soap.

Skin scraping examination was done on the research subjects with potassium hydroxide (KOH) solution to find the mites, alongside pruritus visual analog scale (VAS) score assessment and transepidermal water loss (TEWL) measurement before suitable therapy given. In the first and fourth weeks after the initial assessment, which includes the scabies cure rate, pruritus VAS score, TEWL score, and side effects evaluation, a follow-up was conducted. TEWL was measured using Tewameter® TM 300 made by Courage-Khazaka from Germany. Subsequent data were documented and processed using Statistical Product and Service Product (SPSS) program version 20. Finally, an analysis was done by a third-party which did not seem aware of the treatment given (single-blind).

ELIGIBILITY:
Inclusion Criteria:

* Students diagnosed with scabies and agreed to participate
* Age 12-18 years old
* Has been staying in the boarding school for at least 4 weeks

Exclusion Criteria:

* Not healthy (ie. fever or other conditions which caused subjects were not able to be examined)
* Secondary infection has been found ( yellow crusts, pus, dirty skin lesion, bullae, or systemic symptoms ie. fever)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with scabies a week after first treatment | One week
  Number of participants with scabies a week after first treatment
Number of participants with scabies four weeks after second treatment | Four weeks
  Number of participants with scabies four weeks after second treatment
Transepidermal water loss in gr/hr/m^2 on first week | One week
  Skin barrier damage one week after first treatment
Transepidermal water loss in gr/hr/m^2 on fourth week | Four weeks
  Skin barrier damage one week after second treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Departemen Dermatologi dan Venereologi Fakultas Kedokteran Universitas Indonesia, Jakarta, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No